CLINICAL TRIAL: NCT00333840
Title: A Phase III Study of STI571 Versus Interferon-α (IFN-α) Combined With Cytarabine (Ara-C) in Patients With Newly Diagnosed Previously Untreated Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: Safety and Efficacy of Imatinib Versus Interferon-α Plus Cytarabine in Patients With Newly Diagnosed Philadelphia Chromosome Positive Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571A 0106
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: CML; STI571; imatinib; interferon; interferon alpha; cytosine arabinoside; chronic myeloid leukemia; Philadelphia chromosome positive
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Interferon-alpha; Cytarabine

ARMS (2):
- imatinib (STI571) (Experimental): In the first-line treatment period participants received imatinib 400 mg orally once daily in the morning. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to receive interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 MU/m^2/day. After the maximum tolerated dose of IFN-a was achieved, participants also received cytarabine (ARA-C) 20 mg/m^2/day (max 40 mg) SC injection for 10 days every month. Maximum study duration was 11.5 years.
  Interventions: Drug: imatinib mesilate; Drug: interferon-alpha (INF-a); Drug: cytarabine (ARA-C)
- IFN-a+Ara-C (Active Comparator): In the first-line treatment period participants received interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 MU/m^2/day. After the maximum tolerated dose of IFN-a was achieved, participants also received cytarabine (ARA-C) 20 mg/m^2/day (max 40 mg) SC injections for 10 days every month. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to the second-line treatment period to receive imatinib (STI571). IFN treatment was discontinued with protocol amendment 6. Maximum study duration was 8 years.
  Interventions: Drug: imatinib mesilate; Drug: interferon-alpha (INF-a); Drug: cytarabine (ARA-C)

INTERVENTIONS:
Drug: imatinib mesilate — imatinib supplied as 100 mg and 400 mg tablets or 100 mg capsules.
  Other Names: Glivec®; Gleevec®; STI571
Drug: interferon-alpha (INF-a) — interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 MU/m^2/day.
  Other Names: Roferon®-A; Intron®-A
Drug: cytarabine (ARA-C) — cytarabine 20 mg/m^2/day (max 40 mg) SC for 10 days every month.

SUMMARY:
The purpose of this study is to evaluate and compare the side effects and anti-leukemic benefits of imatinib with those of interferon and Ara-C for patients who have chronic myeloid leukemia (CML) in the chronic phase. Patients in this study will be randomized (1:1) to receive either interferon plus Ara-C or imatinib as initial treatment.

ELIGIBILITY:
Inclusion criteria:

* Must have signed consent for Amendment 5
* Must have completed visit 62 of the core IRIS trial or be in follow-up
* Must be on STI571 treatment
* If on IFN treatment, must be willing to cross over to STI571 treatment

Exclusion criteria:

* Patients who have discontinued from the study and are in follow-up
* Patients who are on IFN treatment and do not want to cross over to STI571 treatment
* Patients who have not consented to amendment 5
* Patients who did not complete the amendment 5 protocol

Additional protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1106 (Actual)
Dates: Start 2000-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (145):
- United States (53):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Montgomery, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Berkeley, California
  - Novartis Investigative Site, Campbell, California
  - Novartis Investigative Site, Duarte, California
  - Novartis Investigative Site, La Jolla, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Honolulu, Hawaii
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Decatur, Illinois
  - Novartis Investigative Site, Beech Grove, Indiana
  - Novartis Investigative Site, Witchita, Kansas
  - Novartis Investigative Site, Louisville, Kentucky
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Detroit, Michigan
  - Novartis Investigative Site, East Lansing, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Billings, Montana
  - Novartis Investigative Site, Omaha, Nebraska
  - Novartis Investigative Site, Hackensack, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Farmington, New Mexico
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Syracuse, New York
  - Novartis Investigative Site, Chapel Hill, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cleveland, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Providence, Rhode Island
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Salt Lake City, Utah
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Milwaukee, Wisconsin
- Australia (11):
  - Novartis Investigative Site, Adelaide
  - Novartis Investigative Site, Brisbane
  - Novartis Investigative Site, Darlinghurst
  - Novartis Investigative Site, East Melbourne
  - Novartis Investigative Site, Nedlands
  - Novartis Investigative Site, Parkville
  - Novartis Investigative Site, Prahan
  - Novartis Investigative Site, South Brisbane
  - Novartis Investigative Site, St Leonards
  - Novartis Investigative Site, Sydney
  - Novartis Investigative Site, Westmead
- Novartis Investigative Site, Vienna, Austria
- Belgium (3):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Godinne
  - Novartis Investigative Site, Leuven
- Canada (10):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Denmark (3):
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Herlev
- France (10):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pessac
  - Novartis Investigative Site, Poitiers
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (15):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Regensburg
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Stuttgart
- Italy (11):
  - Novartis Investigative Site, Bari
  - Novartis Investigative Site, Bologna
  - Novartis Investigative Site, Florence
  - Novartis Investigative Site, Genova
  - Novartis Investigative Site, Milan
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Orbassano
  - Novartis Investigative Site, Pavia
  - Novartis Investigative Site, Pescara
  - Novartis Investigative Site, Pisa
  - Novartis Investigative Site, Reggio Calabria
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Auckland, New Zealand
- Norway (2):
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Tromsø
- Spain (4):
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
  - Novartis Investigative Site, Valencia
- Sweden (7):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Örebro
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Umeå
  - Novartis Investigative Site, Uppsala
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (9):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, Cardiff
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, Liverpool
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Nottingham
  - Novartis Investigative Site, Plymouth

REFERENCES:
- [Derived] Hochhaus A, Larson RA, Guilhot F, Radich JP, Branford S, Hughes TP, Baccarani M, Deininger MW, Cervantes F, Fujihara S, Ortmann CE, Menssen HD, Kantarjian H, O'Brien SG, Druker BJ; IRIS Investigators. Long-Term Outcomes of Imatinib Treatment for Chronic Myeloid Leukemia. N Engl J Med. 2017 Mar 9;376(10):917-927. doi: 10.1056/NEJMoa1609324. PMID 28273028
- [Derived] Jain P, Kantarjian H, Nazha A, O'Brien S, Jabbour E, Romo CG, Pierce S, Cardenas-Turanzas M, Verstovsek S, Borthakur G, Ravandi F, Quintas-Cardama A, Cortes J. Early responses predict better outcomes in patients with newly diagnosed chronic myeloid leukemia: results with four tyrosine kinase inhibitor modalities. Blood. 2013 Jun 13;121(24):4867-74. doi: 10.1182/blood-2013-03-490128. Epub 2013 Apr 25. PMID 23620574
- [Derived] Larson RA, Druker BJ, Guilhot F, O'Brien SG, Riviere GJ, Krahnke T, Gathmann I, Wang Y; IRIS (International Randomized Interferon vs STI571) Study Group. Imatinib pharmacokinetics and its correlation with response and safety in chronic-phase chronic myeloid leukemia: a subanalysis of the IRIS study. Blood. 2008 Apr 15;111(8):4022-8. doi: 10.1182/blood-2007-10-116475. Epub 2008 Feb 6. PMID 18256322

RESULTS

PARTICIPANT FLOW:
Groups:
- Imatinib (STI571): In the first-line treatment period participants received imatinib 400 mg orally once daily in the morning. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to receive interferon-alpha (IFN-a) and cytarabine (ARA-C). Maximum study duration was 11.5 years.
- IFN-a + Ara-C: In the first-line treatment period participants received interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 MU/m^2/day. After the maximum tolerated dose of IFN-a was achieved, participants also received cytarabine (ARA-C) 20 mg/m^2/day (max 40 mg) SC injections for 10 days every month. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to the second-line treatment period to receive imatinib (STI571). IFN treatment was discontinued with protocol amendment 6. Maximum study duration was 8 years.
- Imatinib to IFN-a + Ara-C: In the first-line treatment period participants received imatinib 400 mg orally once daily in the morning. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to receive interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 MU/m^2/day. After the maximum tolerated dose of IFN-a was achieved, participants also received cytarabine (ARA-C) 20 mg/m^2/day (max 40 mg) SC injections for 10 days every month.
- IFN-a + Ara-C to Imatinib: In the first-line treatment period participants received interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 MU/m^2/day. After the maximum tolerated dose of IFN-a was achieved, participants also received cytarabine (ARA-C) 20 mg/m^2/day (max 40 mg) SC injections for 10 days every month. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to the second-line treatment period to receive imatinib (STI571) 400 mg orally once daily in the morning.
Period: First-line Treatment Period
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C | Imatinib to IFN-a + Ara-C | IFN-a + Ara-C to Imatinib
Started | 553 | 553 | 0 | 0
Safety Population; Received Study Drug | 551 | 533 | 0 | 0
Completed | 267 | 7 | 0 | 0
Not Completed | 286 | 546 | 0 | 0
Not completed — Adverse Event | 38 | 37 | 0 | 0
Not completed — Abnormal laboratory values | 3 | 1 | 0 | 0
Not completed — Abnormal procedure | 2 | 0 | 0 | 0
Not completed — Unsatisfactory therapeutic effect | 88 | 29 | 0 | 0
Not completed — No longer required study drug | 21 | 8 | 0 | 0
Not completed — Protocol Violation | 17 | 17 | 0 | 0
Not completed — Subject withdrew consent | 57 | 77 | 0 | 0
Not completed — Lost to Follow-up | 15 | 6 | 0 | 0
Not completed — Administrative problems | 12 | 6 | 0 | 0
Not completed — Death | 19 | 2 | 0 | 0
Not completed — Crossed over to other treatment arm | 14 | 363 | 0 | 0
Period: Second-line Treatment Period
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C | Imatinib to IFN-a + Ara-C | IFN-a + Ara-C to Imatinib
Started | 0 | 0 | 14 | 363
Completed | 0 | 0 | 0 | 175
Not Completed | 0 | 0 | 14 | 188
Not completed — Adverse Event | 0 | 0 | 3 | 34
Not completed — Abnormal Laboratory Values | 0 | 0 | 0 | 3
Not completed — Abnormal procedure | 0 | 0 | 0 | 1
Not completed — Unsatisfactory therapeutic effect | 0 | 0 | 9 | 70
Not completed — No longer required study drug | 0 | 0 | 1 | 14
Not completed — Protocol Violation | 0 | 0 | 1 | 10
Not completed — Subject withdrew consent | 0 | 0 | 0 | 34
Not completed — Lost to Follow-up | 0 | 0 | 0 | 6
Not completed — Administrative problems | 0 | 0 | 0 | 7
Not completed — Death | 0 | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- IFN-a + Ara-C: In the first-line treatment period participants received interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 MU/m^2/day. After the maximum tolerated dose of IFN-a was achieved, participants also received cytarabine (ARA-C) 20 mg/m^2/day (max 40 mg) SC injections for 10 days every month. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to the second-line treatment period to receive imatinib (CSI151). IFN treatment was discontinued with protocol amendment 6. Maximum study duration was 8 years.
- Total: Total of all reporting groups
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C | Total
Number analyzed (Participants) | 553 | 553 | 1106
Age Continuous [Median (Full Range); unit: years] | 50.0 [18 to 70] | 51.0 [18 to 70] | 51.0 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 243 | 454
  Male | 342 | 310 | 652

OUTCOME MEASURES:

1. Primary Outcome: Kaplan-Meier Estimates of Overall Survival (All Randomized Participants)
Description: Overall survival was defined as the time between date of randomization and death due to any cause. The time was censored at last examination date for patients who were still being treated and at date of last contact for patients who discontinued treatment. Kaplan-Meier estimates of the percentage of participants at each time point was calculated. This outcome was measured in all randomized patients, regardless of whether crossover occurred, i.e., events that occurred in patients, who had crossed over, were attributed following crossover to the original randomized treatment.
Time Frame: 12,24,36,48,60,72,84,96,108,120,132 and 144 months
Population: Intent-to-treat population included all randomized participants. n = number of participants at risk at the beginning of the specific time interval
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C
Number analyzed (Participants) | 553 | 553
Percentage of participants
  12 months (n = 553, 553) | 98.9 [98 to 100] | 97.7 [96 to 99]
  24 months (n = 542, 512) | 96.0 | 93.6
  36 months (n = 518, 471) | 92.4 | 89.8
  48 months (n = 492, 441) | 90.4 | 87.7
  60 months (n = 475, 411) | 89.4 | 85.4
  72 months (n = 461, 388) | 88.2 | 83.8
  84 months (n = 446, 373) | 86.6 | 83.1
  96 months (n = 430, 358) | 85.4 | 81.4
  108 months (n = 391, 315) | 84.3 | 79.9
  120 months (n = 368, 299) | 83.3 | 78.8
  132 months (n = 356, 288) | 82.8 | 77.7
  144 months (n = 250, 199) | 81.3 | 75.4

2. Secondary Outcome: Kaplan Meier Estimates of Event Free Survival (All Randomized Participants)
Description: Event-free survival is defined as the time between randomization and the earliest of any of the following events on treatment:
  * progression to Accelerated Phase (AP) or Blast Crisis (BC)
  * loss of Complete Hematological Response (CHR)
  * loss of Major Cytogenetic Response (MCyR) confirmed
  * loss of Major Cytogenetic Response (MCyR) unconfirmed
  * increase in white blood cell count (WBC) if approved by the Study Management Committee (SMC)
  * death (due to any cause when reported as primary reason for discontinuation of treatment).
  Kaplan Meier estimates of the percentage of participants with Event Free Survival at the given time point was calculated. This outcome was measured in all randomized patients, regardless of whether crossover occurred, i.e., events that occurred in patients, who had crossed over, were attributed following crossover to the original randomized treatment.
Time Frame: 12,24,36,48,60,72,84,96,108,120,132 and 144 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C
Number analyzed (Participants) | 553 | 553
Percentage of participants
  12 months (n = 553, 553) | 96.6 | 79.4
  24 months (n = 505, 332) | 89.6 | 70.0
  36 months (n = 448, 263) | 85.3 | 67.0
  48 months (n = 415, 241) | 83.9 | 63.7
  60 months (n = 395, 223) | 83.2 | 61.9
  72 months (n = 376, 207) | 83.0 | 60.1
  84 months (n = 352, 181) | 82.0 | 59.0
  96 months (n = 334, 166) | 81.0 | 58.3
  108 months (n = 301, 141) | 79.9 | 56.6
  120 months (n = 269, 130) | 79.6 | 56.6
  132 months (n = 257, 124) | 79.6 | 56.6
  144 months (n = 143, 76) | 79.6 | 51.8

3. Secondary Outcome: Percentage of Participants With Event Free Survival Events (All Randomized Participants)
Description: Event-free survival is defined as the time between randomization and the earliest of any of the following events on treatment:
  * progression to Accelerated Phase (AP) or Blast Crisis (BC)
  * loss of Complete Hematological Response (CHR)
  * loss of Major Cytogenic Response (MCyR) confirmed
  * loss of Major Cytogenic Response (MCyR) unconfirmed
  * increase in white blood cell count (WBC) if approved by the Study Management Committee (SMC)
  * death (due to any cause when reported as primary reason for discontinuation of treatment).
  The percentage of participants with Event Free Survival events in each category was calculated. This outcome was measured in all randomized patients, regardless of whether crossover occurred, i.e., events that occurred in patients, who had crossed over, were attributed following crossover to the original randomized treatment.
Time Frame: 144 months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C
Number analyzed (Participants) | 553 | 553
Percentage of participants
  Participants with events | 17.9 | 32.2
  Progression to AP or BC | 6.9 | 12.8
  Loss of CHR | 2.7 | 7.6
  Loss of MCyR (confirmed) | 4.2 | 5.4
  Loss of MCyR (unconfirmed) | 0.9 | 1.1
  Increase of WBC | 0.2 | 3.4
  Death | 3.1 | 1.8

4. Secondary Outcome: Kaplan Meier Estimates of Time to Progression to Accelerated Phase (AP) or Blast Crisis (BC) (All Randomized Participants)
Description: Time to progression to AP/BC is defined as the time between randomization and either of the following events on treatment: death (due to CML when reported as primary reason for discontinuation of treatment) or progression to Accelerated Phase or Blast Crisis and is censored at last examination date for patients without event. No data after discontinuation of study treatment was included. The Kaplan Meier estimates of the percentage of participants with survival without progression to AP/BC at the given time point was calculated. This outcome was measured in all randomized patients, regardless of whether crossover occurred, i.e., events that occurred in patients, who had crossed over, were attributed following crossover to the original randomized treatment.
Time Frame: 12,24,36,48,60,72,84,96,108,120,132 and 144 months
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Groups:
- Imatinib (STI571): In the first-line treatment period participants received imatinib 400 mg orally once daily in the morning. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to receive interferon-alpha (IFN-a) and cytarabine (ARA-C) in the second-line treatment period. Maximum study duration was 11.5 years.
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C
Number analyzed (Participants) | 553 | 553
Percentage of participants
  12 months (n = 553, 553) | 98.5 | 92.9
  24 months (n = 513, 388) | 95.7 | 90.0
  36 months (n = 461, 337) | 94.0 | 87.9
  48 months (n = 431, 311) | 93.1 | 84.7
  60 months (n = 409, 289 ) | 92.7 | 83.5
  72 months (n = 384, 265) | 92.7 | 83.1
  84 months (n = 358, 236) | 92.7 | 82.4
  96 months (n = 338, 220) | 92.4 | 82.4
  108 months (n = 305, 189) | 92.1 | 82.4
  120 months (n = 272, 175) | 92.1 | 82.4
  132 months (n = 259, 165) | 92.1 | 82.4
  144 months (n = 145, 94) | 92.1 | 82.4

5. Secondary Outcome: Percentage of Participants With Best Cytogenetic Response (First-line Treatment)
Description: Bone marrow aspirate was performed to evaluate cytogenetic results (percentage of Philadelphia chromosome positive (Ph+) metaphases) and amount of blasts and promyelocytes in bone marrow to establish cytogenetic response.
  Major Cytogenetic Response= Complete Response or Partial Response. Complete Cytogenetic Response= 0 % of Ph+ metaphases (out of 20 metaphases). Partial Cytogenetic Response= > 0 and ≤ 35 % of Ph+ metaphases (out of 20 metaphases). The percentage of participants with cytogenetic response in each category was calculated.
Time Frame: 144 months
Population: Intent-to-treat participants included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C
Number analyzed (Participants) | 553 | 553
Percentage of participants
  Major Cytogenic Response | 89.0 | 23.3
  Complete Cytogenic Response | 82.8 | 11.6
  Partial Cytogenic Response | 6.1 | 11.8

6. Secondary Outcome: Percentage of Participants With Best Cytogenetic Response (Second-line Treatment)
Description: Bone marrow aspirate was performed to evaluate cytogenetic results (percentage of Ph chromosome (Ph+) containing metaphases) and the amount of blasts and promyelocytes in bone marrow to establish cytogenetic response.
  Major Cytogenetic Response= Complete Response or Partial Response. Complete Cytogenetic Response= 0 % of Ph+ metaphases (out of 20 metaphases). Partial Cytogenetic Response= > 0 and ≤ 35 % Ph+ metaphases (out of 20 metaphases). The percentage of participants with cytogenetic response in each category was calculated.
Time Frame: 144 months
Population: Intent-to-treat participants included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib to IFN-a + Ara-C | IFN-a + Ara-C to Imatinib
Number analyzed (Participants) | 14 | 363
Percentage of participants
  Major Cytogenic Response | 14.3 | 86.0
  Complete Cytogenic Response | 7.1 | 81.0
  Partial Cytogenic Response | 7.1 | 5.0

7. Secondary Outcome: Number of Participants With Serious Adverse Events as a Measure of Safety (First-line Treatment)
Description: A serious adverse event is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, requires in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant
Time Frame: 144 months
Population: Safety Population included all randomized participants who received study drug.
Measure: Number; unit: Participants
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C
Number analyzed (Participants) | 551 | 533
Participants | 226 | 163

8. Secondary Outcome: Number of Participants With Serious Adverse Events as a Measure of Safety (Second-line Treatment)
Description: as for outcome 7
Time Frame: 144 months
Population: Safety Population included all randomized participants who received study drug.
Measure: Number; unit: Participants
Groups:
- Imatinib to IFN-a + Ara-C: In the first-line treatment period participants received imatinib 400 mg orally once daily in the morning. Hydroxyurea was permitted in the first 6 months to keep the white blood cell count (WBC) below 20.0 X 10^9/liter. If protocol specific criteria applied, participants were eligible to crossover to receive interferon-alpha (IFN-a) subcutaneous (SC) injections escalated over 4 weeks to achieve a target dose of 5 mu/m^2/day. After the maximum tolerated dose of IFN-a was achieved, participants also received cytarabine (ARA-C) 20 mg/m^2/day (max 40 mg) SC injection for 10 days every month in the second-line treatment period.
Arm/Group | Imatinib to IFN-a + Ara-C | IFN-a + Ara-C to Imatinib
Number analyzed (Participants) | 14 | 363
Participants | 2 | 160

9. Secondary Outcome: Percentage of Participants With Major Molecular Response (First-line Treatment)
Description: Major Molecular Response was determined using a quantitative polymerase chain reaction (PCR) laboratory test and was defined as BCR-ABL protein transcripts of ≤ 0.1% according to the international scale.
Time Frame: 12,24,36,48,60,72,84,96,108,120,132 and 144 months
Population: Intent-to-treat population included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C
Number analyzed (Participants) | 553 | 553
Percentage of participants
  12 months (n= 305, 83) | 50.2 | 9.6
  24 months (n= 102, 12) | 69.6 | 25.0
  36 months (n= 68, 7) | 76.5 | 28.6
  48 months (n= 305, 12) | 77.0 | 58.3
  60 months (n= 316, 10) | 88.0 | 100.0
  72 months (n= 292, 9) | 88.0 | 88.9
  84 months (n= 247, 8) | 91.9 | 87.5
  96 months (n= 228, 4) | 92.5 | 100.0
  108 months (n= 233, 0) | 93.6 | NA — Because this table refers to first-line therapy only and not cross-over, no participants were available for testing from Month 108 to Month 144.
  120 months (n= 204, 0) | 93.1 | NA — Because this table refers to first-line therapy only and not cross-over, no participants were available for testing from Month 108 to Month 144.
  132 months (n= 168, 0) | 92.3 | NA — Because this table refers to first-line therapy only and not cross-over, no participants were available for testing from Month 108 to Month 144.
  144 months (n= 1, 0) | 100.0 | NA — Because this table refers to first-line therapy only and not cross-over, no participants were available for testing from Month 108 to Month 144.

10. Secondary Outcome: Percentage of Participants With Major Molecular Response (Second-line Treatment)
Description: as for outcome 9
Time Frame: 12,24,36,48,60,72,84,96,108,120,132 and 144 months
Population: Intent-to-treat population included all randomized participants. No participants in the imatinib to IFN-a + Ara-C arm were available for testing.
Measure: Number; unit: Percentage of participants
Arm/Group | IFN-a + Ara-C to Imatinib
Number analyzed (Participants) | 363
Percentage of participants
  12 months (n = 86) | 51.2
  24 months (n = 62) | 69.4
  36 months (n = 130) | 78.5
  48 months (n = 216) | 81.9
  60 months (n = 174) | 86.2
  72 months (n = 146) | 91.1
  84 months (n = 139) | 86.3
  96 months (n = 138) | 87.0
  108 months (n = 120) | 90.0
  120 months (n = 84) | 85.7
  132 months (n = 31) | 90.3
  144 months | NA — No participants were available for testing at this specific time point, or patients had no PCR assessment done.

ADVERSE EVENTS:
Arm/Group | Imatinib (STI571) | IFN-a + Ara-C | Imatinib to IFN-a + Ara-C | IFN-a + Ara-C to Imatinib
Serious Adverse Events (participants affected / at risk) | 226/551 | 163/533 | 2/14 | 160/363
Other Adverse Events (participants affected / at risk) | 541/551 | 531/533 | 13/14 | 347/363
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (STI571) (N=551) | IFN-a + Ara-C (N=533) | Imatinib to IFN-a + Ara-C (N=14) | IFN-a + Ara-C to Imatinib (N=363)
Acquired Von Willebrand's disease (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 10 | 0 | 5
Autoimmune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Haematotoxicity (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Haemolysis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 4
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 10 | 0 | 1
Thrombocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 2
Angina pectoris (Cardiac disorders) | 2 | 1 | 0 | 2
Angina unstable (Cardiac disorders) | 1 | 1 | 0 | 0
Aortic valve disease (Cardiac disorders) | 0 | 0 | 0 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 4 | 1 | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 3 | 0 | 3
Bradycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 5 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 2 | 0 | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 4 | 4 | 0 | 2
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0 | 1
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0 | 0
Conduction disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 7 | 1 | 0 | 2
Heart valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1 | 0 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 2 | 1 | 0 | 3
Left ventricular failure (Cardiac disorders) | 0 | 0 | 0 | 1
Mitral valve stenosis (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 7 | 5 | 0 | 2
Nodal arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Torsade de pointes (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0
Gene mutation (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Sensory neuropathy hereditary (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Goitre (Endocrine disorders) | 1 | 0 | 0 | 2
Hyperparathyroidism (Endocrine disorders) | 0 | 0 | 0 | 1
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Blindness (Eye disorders) | 0 | 1 | 0 | 0
Blindness unilateral (Eye disorders) | 1 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 2 | 0 | 0 | 0
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0 | 0
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 2 | 0 | 0 | 0
Open angle glaucoma (Eye disorders) | 1 | 0 | 0 | 0
Papilloedema (Eye disorders) | 1 | 0 | 0 | 0
Retinal detachment (Eye disorders) | 1 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 1 | 1 | 0 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 1 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 12 | 1 | 0 | 5
Abdominal pain lower (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3 | 0 | 2
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Acute abdomen (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Crohn's disease (Gastrointestinal disorders) | 3 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 9 | 2 | 0 | 5
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticular perforation (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Duodenitis (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Faecal vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 3
Gastritis erosive (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 0 | 0 | 2
Gastrointestinal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 2 | 2 | 0 | 2
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 7 | 8 | 0 | 4
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Painful defaecation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 3 | 2 | 0 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 2 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Vomiting (Gastrointestinal disorders) | 11 | 7 | 0 | 2
Abasia (General disorders) | 1 | 0 | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 4 | 0 | 3
Cardiac death (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 1 | 1 | 0 | 1
Chest pain (General disorders) | 14 | 4 | 0 | 7
Chills (General disorders) | 7 | 4 | 0 | 1
Condition aggravated (General disorders) | 0 | 0 | 0 | 1
Crepitations (General disorders) | 1 | 0 | 0 | 0
Device malfunction (General disorders) | 1 | 0 | 0 | 0
Drug ineffective (General disorders) | 1 | 1 | 0 | 2
Drug interaction (General disorders) | 1 | 0 | 0 | 0
Drug intolerance (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 3 | 7 | 1 | 3
Gait disturbance (General disorders) | 0 | 1 | 0 | 0
General physical health deterioration (General disorders) | 0 | 2 | 0 | 3
Generalised oedema (General disorders) | 0 | 0 | 0 | 1
Granuloma (General disorders) | 1 | 0 | 0 | 0
Hernia (General disorders) | 1 | 0 | 0 | 0
Hyperplasia (General disorders) | 0 | 0 | 0 | 1
Hyperthermia (General disorders) | 0 | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 2 | 0 | 0 | 1
Malaise (General disorders) | 4 | 2 | 0 | 0
Mucosal atrophy (General disorders) | 0 | 0 | 0 | 1
Multi-organ failure (General disorders) | 1 | 0 | 0 | 0
Necrosis (General disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 3 | 1 | 0 | 0
Pain (General disorders) | 4 | 1 | 0 | 1
Performance status decreased (General disorders) | 1 | 2 | 0 | 1
Pyrexia (General disorders) | 19 | 20 | 1 | 12
Soft tissue inflammation (General disorders) | 1 | 0 | 0 | 0
Spinal pain (General disorders) | 1 | 0 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Biliary tract disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 6 | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 4 | 2 | 0 | 2
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Granulomatous liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1 | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0
Transplant rejection (Immune system disorders) | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 2 | 0 | 0 | 1
Amoebiasis (Infections and infestations) | 0 | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 4 | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bone tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 6 | 3 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 3 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1
Gastritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 0 | 3
Gastroenteritis norovirus (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 0
Haemophilus infection (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 1
Incision site infection (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 2
Influenza (Infections and infestations) | 1 | 0 | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2
Lung infection (Infections and infestations) | 1 | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 1 | 0 | 0 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Meningoencephalitis herpetic (Infections and infestations) | 0 | 0 | 0 | 1
Muscle abscess (Infections and infestations) | 1 | 1 | 0 | 0
Mycoplasma infection (Infections and infestations) | 0 | 1 | 0 | 0
Necrotising fasciitis (Infections and infestations) | 0 | 1 | 0 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Orchitis (Infections and infestations) | 0 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Pelvic abscess (Infections and infestations) | 2 | 0 | 0 | 0
Peridiverticular abscess (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 12 | 7 | 0 | 14
Pneumonia streptococcal (Infections and infestations) | 0 | 0 | 0 | 1
Post procedural infection (Infections and infestations) | 1 | 1 | 0 | 0
Prostate infection (Infections and infestations) | 0 | 0 | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2 | 0 | 0
Rectal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 0 | 2
Salpingitis (Infections and infestations) | 0 | 1 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Scrotal gangrene (Infections and infestations) | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 3 | 1 | 0 | 2
Septic shock (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 2 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 2 | 1 | 0 | 0
Streptococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Systemic candida (Infections and infestations) | 0 | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 2 | 0 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Tuberculoma of central nervous system (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 4 | 4 | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 1
Viral infection (Infections and infestations) | 3 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vulvitis (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Exposure via father (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Graft dysfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Meniscus lesion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Skull fractured base (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Urethral stricture postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Vascular injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 1 | 0 | 1
Amylase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase abnormal (Investigations) | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 1
Blast cell count increased (Investigations) | 0 | 0 | 0 | 1
Blast cells present (Investigations) | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine increased (Investigations) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 1
Blood culture positive (Investigations) | 1 | 0 | 0 | 0
Blood parathyroid hormone increased (Investigations) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Body temperature increased (Investigations) | 1 | 1 | 0 | 0
Creatinine renal clearance decreased (Investigations) | 1 | 0 | 0 | 0
Echocardiogram abnormal (Investigations) | 0 | 1 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 2
Heart rate increased (Investigations) | 0 | 0 | 0 | 1
Hepatic enzyme increased (Investigations) | 2 | 0 | 0 | 0
Lipase increased (Investigations) | 2 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 2
Multiple gated acquisition scan abnormal (Investigations) | 0 | 0 | 0 | 1
Myelocyte present (Investigations) | 0 | 0 | 0 | 1
Platelet count increased (Investigations) | 0 | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0 | 1
Troponin increased (Investigations) | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 2 | 1 | 0 | 2
White blood cell count increased (Investigations) | 0 | 4 | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 3 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 5 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Food intolerance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 11 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 6 | 0 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 6 | 1 | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Inclusion body myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 3
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 10 | 0 | 2
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 0 | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Acral lentiginous melanoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 3
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0 | 1
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Blast cell crisis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Blast crisis in myelogenous leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5 | 0 | 12
Bone neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1 | 0 | 3
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Carcinoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chloroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Chronic lymphocytic leukaemia transformation (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 3
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Erythroleukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lip and/or oral cavity cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 1
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastases to adrenals (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to large intestine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 2
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0 | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 1 | 3
Neoplasm of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 1 | 0 | 9
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0 | 0
Signet-ring cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 0 | 1
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 0 | 0 | 1
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Areflexia (Nervous system disorders) | 1 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 1 | 3 | 0 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Brain mass (Nervous system disorders) | 0 | 0 | 0 | 1
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2 | 0 | 2
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Coma (Nervous system disorders) | 1 | 0 | 0 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Complicated migraine (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 1
Dementia (Nervous system disorders) | 0 | 2 | 0 | 0
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1 | 0 | 0
Demyelination (Nervous system disorders) | 1 | 0 | 0 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 7 | 5 | 1 | 0
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 2 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 3 | 3 | 0 | 2
Hemiparesis (Nervous system disorders) | 1 | 1 | 0 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 1 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 1 | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 2 | 0 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Multiple sclerosis (Nervous system disorders) | 1 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Paraplegia (Nervous system disorders) | 0 | 1 | 0 | 0
Parkinson's disease (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 0 | 1
Piriformis syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Polyneuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 1 | 0 | 0
Radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 2 | 0 | 0
Simple partial seizures (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0
Speech disorder (Nervous system disorders) | 0 | 2 | 0 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 8 | 4 | 0 | 2
Temporal lobe epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Transient global amnesia (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 3 | 0 | 3
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Aggression (Psychiatric disorders) | 0 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 2 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 3 | 0 | 0
Completed suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 3 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 2 | 15 | 0 | 2
Depression suicidal (Psychiatric disorders) | 0 | 2 | 0 | 0
Disorientation (Psychiatric disorders) | 0 | 1 | 0 | 0
Homicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 0
Mania (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0
Paranoia (Psychiatric disorders) | 0 | 0 | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 5 | 0 | 0
Acute prerenal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0
Calculus ureteric (Renal and urinary disorders) | 0 | 1 | 0 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 6 | 0 | 0 | 1
Nephrotic syndrome (Renal and urinary disorders) | 0 | 1 | 0 | 0
Oliguria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 5 | 2 | 0 | 3
Renal failure acute (Renal and urinary disorders) | 5 | 0 | 0 | 2
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 1 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 2 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 1 | 0 | 2
Penis disorder (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Prostatic dysplasia (Reproductive system and breast disorders) | 2 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Testicular swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vaginal cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Varicose veins pelvic (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 0 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 3
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Polymorphic light eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Cardiac assistance device user (Social circumstances) | 0 | 1 | 0 | 0
Disability (Social circumstances) | 0 | 1 | 0 | 0
Miscarriage of partner (Social circumstances) | 1 | 0 | 0 | 0
Abortion induced (Surgical and medical procedures) | 1 | 0 | 0 | 1
Abscess drainage (Surgical and medical procedures) | 1 | 0 | 0 | 0
Bone marrow transplant (Surgical and medical procedures) | 0 | 0 | 0 | 1
Coronary arterial stent insertion (Surgical and medical procedures) | 0 | 0 | 0 | 1
Stem cell transplant (Surgical and medical procedures) | 0 | 0 | 0 | 1
Aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Arterial occlusive disease (Vascular disorders) | 2 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 2 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 2 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0 | 1
Femoral artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0
Haemorrhage (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 4 | 0 | 0
Iliac artery occlusion (Vascular disorders) | 1 | 0 | 0 | 0
Iliac artery stenosis (Vascular disorders) | 1 | 0 | 0 | 0
Infarction (Vascular disorders) | 1 | 0 | 0 | 0
Ischaemia (Vascular disorders) | 0 | 0 | 0 | 3
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Varicophlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Vascular occlusion (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Imatinib (STI571) (N=551) | IFN-a + Ara-C (N=533) | Imatinib to IFN-a + Ara-C (N=14) | IFN-a + Ara-C to Imatinib (N=363)
Anaemia (Blood and lymphatic system disorders) | 64 | 58 | 0 | 37
Leukopenia (Blood and lymphatic system disorders) | 26 | 28 | 2 | 14
Monocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 58 | 68 | 1 | 56
Pancytopenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 70 | 129 | 4 | 44
Thrombocytosis (Blood and lymphatic system disorders) | 7 | 3 | 1 | 6
Deafness (Ear and labyrinth disorders) | 2 | 5 | 1 | 3
Ear pain (Ear and labyrinth disorders) | 17 | 18 | 1 | 8
Vertigo (Ear and labyrinth disorders) | 22 | 39 | 0 | 16
Hypothyroidism (Endocrine disorders) | 3 | 11 | 1 | 3
Conjunctivitis (Eye disorders) | 46 | 27 | 0 | 21
Dry eye (Eye disorders) | 20 | 16 | 1 | 11
Eye pain (Eye disorders) | 14 | 23 | 1 | 7
Eye swelling (Eye disorders) | 50 | 7 | 0 | 19
Eyelid oedema (Eye disorders) | 49 | 7 | 0 | 29
Growth of eyelashes (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation increased (Eye disorders) | 42 | 4 | 0 | 15
Periorbital oedema (Eye disorders) | 165 | 6 | 0 | 98
Retinal exudates (Eye disorders) | 0 | 2 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 40 | 10 | 0 | 16
Abdominal pain (Gastrointestinal disorders) | 90 | 62 | 1 | 56
Abdominal pain upper (Gastrointestinal disorders) | 74 | 64 | 0 | 38
Constipation (Gastrointestinal disorders) | 63 | 77 | 2 | 27
Diarrhoea (Gastrointestinal disorders) | 250 | 231 | 2 | 148
Dry mouth (Gastrointestinal disorders) | 16 | 58 | 1 | 9
Dyspepsia (Gastrointestinal disorders) | 105 | 44 | 1 | 53
Flatulence (Gastrointestinal disorders) | 40 | 8 | 0 | 16
Gastric disorder (Gastrointestinal disorders) | 3 | 3 | 1 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 35 | 13 | 0 | 21
Gingival bleeding (Gastrointestinal disorders) | 5 | 19 | 1 | 3
Haemorrhoids (Gastrointestinal disorders) | 19 | 12 | 1 | 6
Mouth ulceration (Gastrointestinal disorders) | 7 | 33 | 1 | 9
Nausea (Gastrointestinal disorders) | 276 | 325 | 4 | 138
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 11 | 55 | 0 | 6
Vomiting (Gastrointestinal disorders) | 126 | 145 | 2 | 68
Asthenia (General disorders) | 43 | 87 | 2 | 30
Chest pain (General disorders) | 46 | 47 | 0 | 20
Chills (General disorders) | 47 | 179 | 3 | 19
Fatigue (General disorders) | 214 | 354 | 7 | 104
Influenza like illness (General disorders) | 38 | 85 | 3 | 17
Local swelling (General disorders) | 6 | 1 | 2 | 3
Malaise (General disorders) | 7 | 41 | 0 | 6
Mucosal inflammation (General disorders) | 6 | 55 | 0 | 5
Oedema (General disorders) | 46 | 6 | 0 | 37
Oedema peripheral (General disorders) | 134 | 31 | 0 | 94
Pain (General disorders) | 29 | 52 | 0 | 14
Pyrexia (General disorders) | 91 | 217 | 3 | 42
Cholestasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 5 | 15 | 1 | 11
Bronchitis (Infections and infestations) | 54 | 40 | 0 | 34
Cystitis (Infections and infestations) | 13 | 7 | 1 | 10
Gastroenteritis (Infections and infestations) | 35 | 9 | 0 | 12
Influenza (Infections and infestations) | 77 | 33 | 0 | 29
Nasopharyngitis (Infections and infestations) | 167 | 47 | 2 | 84
Pharyngitis (Infections and infestations) | 23 | 24 | 1 | 11
Rhinitis (Infections and infestations) | 42 | 18 | 0 | 14
Sinusitis (Infections and infestations) | 63 | 32 | 2 | 29
Upper respiratory tract infection (Infections and infestations) | 114 | 45 | 0 | 50
Urinary tract infection (Infections and infestations) | 36 | 31 | 0 | 26
Animal bite (Injury, poisoning and procedural complications) | 3 | 1 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 30 | 15 | 0 | 14
Muscle injury (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0
Alanine aminotransferase abnormal (Investigations) | 1 | 3 | 1 | 2
Alanine aminotransferase increased (Investigations) | 24 | 31 | 1 | 11
Haemoglobin decreased (Investigations) | 11 | 9 | 1 | 9
Platelet count decreased (Investigations) | 4 | 8 | 1 | 8
Weight decreased (Investigations) | 26 | 91 | 1 | 14
Weight increased (Investigations) | 86 | 14 | 1 | 52
White blood cell count increased (Investigations) | 3 | 8 | 1 | 3
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 53 | 207 | 2 | 18
Dehydration (Metabolism and nutrition disorders) | 7 | 11 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 29 | 3 | 0 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 37 | 12 | 0 | 22
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 173 | 199 | 3 | 93
Back pain (Musculoskeletal and connective tissue disorders) | 137 | 105 | 2 | 59
Bone pain (Musculoskeletal and connective tissue disorders) | 58 | 78 | 2 | 28
Muscle spasms (Musculoskeletal and connective tissue disorders) | 272 | 63 | 1 | 168
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 34 | 30 | 1 | 19
Myalgia (Musculoskeletal and connective tissue disorders) | 131 | 200 | 4 | 63
Neck pain (Musculoskeletal and connective tissue disorders) | 26 | 11 | 1 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 107 | 89 | 0 | 53
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 1 | 1
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1 | 2
Ageusia (Nervous system disorders) | 1 | 4 | 1 | 0
Amnesia (Nervous system disorders) | 10 | 35 | 0 | 9
Disturbance in attention (Nervous system disorders) | 7 | 37 | 1 | 3
Dizziness (Nervous system disorders) | 105 | 124 | 3 | 43
Dizziness postural (Nervous system disorders) | 0 | 3 | 1 | 2
Dysarthria (Nervous system disorders) | 0 | 2 | 1 | 0
Dysgeusia (Nervous system disorders) | 17 | 48 | 1 | 8
Headache (Nervous system disorders) | 205 | 231 | 2 | 87
Lethargy (Nervous system disorders) | 11 | 36 | 0 | 3
Memory impairment (Nervous system disorders) | 4 | 9 | 1 | 3
Migraine (Nervous system disorders) | 14 | 6 | 1 | 7
Neuropathy peripheral (Nervous system disorders) | 14 | 24 | 1 | 11
Paraesthesia (Nervous system disorders) | 50 | 39 | 0 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 4 | 3 | 1 | 0
Anxiety (Psychiatric disorders) | 52 | 60 | 3 | 17
Depression (Psychiatric disorders) | 84 | 186 | 3 | 31
Disorientation (Psychiatric disorders) | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 83 | 99 | 0 | 31
Mood altered (Psychiatric disorders) | 3 | 22 | 1 | 2
Nervousness (Psychiatric disorders) | 9 | 7 | 1 | 6
Dysuria (Renal and urinary disorders) | 11 | 15 | 2 | 5
Polyuria (Renal and urinary disorders) | 2 | 2 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 3 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 111 | 122 | 4 | 54
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2 | 7 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 50 | 75 | 1 | 33
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 | 42 | 0 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 100 | 61 | 3 | 25
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 | 20 | 1 | 7
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 30 | 125 | 2 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 46 | 44 | 1 | 20
Erythema (Skin and subcutaneous tissue disorders) | 40 | 23 | 0 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 33 | 79 | 0 | 20
Night sweats (Skin and subcutaneous tissue disorders) | 55 | 84 | 2 | 27
Pruritus (Skin and subcutaneous tissue disorders) | 53 | 63 | 0 | 24
Rash (Skin and subcutaneous tissue disorders) | 154 | 91 | 0 | 78
Haematoma (Vascular disorders) | 9 | 8 | 2 | 6
Hypertension (Vascular disorders) | 50 | 16 | 0 | 23
Peripheral coldness (Vascular disorders) | 4 | 7 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.